CLINICAL TRIAL: NCT05909384
Title: Expert Consensus Statements for the Management of Sepsis in Resource Limited Settings Using a Delphi Method
Brief Title: Management of Sepsis in Resource Limited Settings Using a Delphi Method.
Status: Completed | Type: Observational
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Asia Pacific Sepsis Alliance (Unknown)
Responsible Party: Sponsor
Other Study IDs: APSADelphi_V1.2
Record Dates: First submitted 2023-05-19; First posted 2023-06-18 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Sepsis
Keywords: Sepsis; Septic shock; Low- and middle- income countries; LMIC; Delphi; Resource-limited setting
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert group: 1. Clinical expertise in adult sepsis management, AND
  2. Demonstrated involvement with sepsis related research, educations, policy/protocols, professional activities
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Multiple rounds of surveys collecting information on sepsis diagnosis and management in resource-limited settings.

SUMMARY:
Rapid evolution of sepsis syndromes means that timely diagnosis and treatment are critical in improving outcomes but this may be difficult to achieve in many low- and middle- income countries (LMICs) and there is a lack of high quality clinical evidence to guide diagnosis and management in LMIC settings. The wide variability in health systems in LMICs means that additional areas of guidance may be required where staff or facilities are lacking. In the absence of clinical data, to address some of these issues, the investigators aim to use Delphi methodology to obtain experts consensus statements on some specific aspects of sepsis management in LMICs.

DETAILED DESCRIPTION:
The investigators aim to use a Delphi process to generate expert consensus practice statements in the context of diagnosis and management of sepsis in LMICs, including identification of aspects of sepsis diagnosis and management in LMICs not covered by existing guidelines. The questions will undergo several iterative rounds and will be in multiple-choice or Likert scale format. A study steering group will review the results of each round via video conference and design the questionnaire for the next survey. Summary results of each round will be presented to experts, along with the survey questionnaire for the next round. The survey process will be repeated with the modified questionnaire. The Delphi rounds will continue until the desired consensus and stability are achieved.

ELIGIBILITY:
Inclusion Criteria:

* Recognized experts meeting pre-defined criteria (below) from a wide geographical distribution with approximately 70% from LMICs.

  1. Clinical expertise in adult sepsis management, AND
  2. Demonstrated involvement with sepsis related research, educations, policy/protocols, professional activities

     Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recognized experts meeting pre-defined criteria from a wide geographical distribution with approximately 70% from LMICs
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire statements which have reached pre-defined consensus | 2 weeks
  Descriptive analysis of questionnaire statements which have reached pre-defined consensus. Consensus will be defined as >70% participants in favour of agree/disagree statements (Likert scale 1-3 means disagree or 5-7 means agree), or >80% in favour of single option in a single stem question with multiple responses (yes/no answers).

CONTACTS AND LOCATIONS:
Overall Officials: Brett Abbenbroek, BSc,MPH,PhD, Study Director — The George Institute
Locations (1):
- Oxford University Clinical Research Unit, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No